CLINICAL TRIAL: NCT05138692
Title: The Association Between Initial Concentrations of Biomarkers and Outcome 1 and 10-15 Years After Severe Traumatic Brain Injury
Brief Title: Biomarkers and Outcome 1 and 10-15 Years After Severe Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Bengt Nellgard (Other)
Collaborators: Svenska alzheimerfonden (Unknown); Stroke Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Bengt Nellgard, Associate professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Other Study IDs: Neuromarkers and neurotrauma
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Brain Injury Traumatic Severe (Diagnosis); Biomarkers
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Biomarkers Neurofilament light (NFL) and Glial Fibrillary Acid Protein (GFAP) were analyzed in CSF, TAU in serum, APOE- genotype was explored in whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After written consent from next-of-kin patients with severe traumatic brain injury was included from the neurointensive care unit (NICU) at Sahlgrenska university hospital, Gothenburg. Blood and CSF samples were collected during the initial 3 weeks after trauma. 1 year after trauma patients were assessed according to Glasgow outcome scale (GOS), NIHSS and Barthels. 10-15 years after trauma a repeated evaluation according to GOS was performed by telephone. Different biomarkers such as Neurofilament light, Glial fibrillary acidic protein and Tau among others, was analyzed from serum and CSF samples. Further patients were explored Apolipoprotein-E genetype (APOE). The investigators hypothesize that higher biomarkers concentrations and positive test for this gene relate to worse outcome 1-year and 10-15 years after trauma. Further that these biomarkers and genetic marker further have prognostic value on outcome 1-year and 10-15 years after trauma. Finally, the investigators want to explore the concentrations dynamics of these biomarkers in serum and CSF in the acute phase after trauma.

DETAILED DESCRIPTION:
Patients with a severe traumatic brain injury (sTBI) were included after written consent from next-to kin. The injury was considered as severe if having a Glasgow coma scale of 8 or less. Within 48h of trauma patients were included from the neurointensive care unit at Sahlgrenska university hospital, Gothenburg during 2000-2004. Patients were intubated and had a ventricular catheter. All patients were treated in accordance with the Lund Concept. Samples from ventricular cerebrospinal fluid (CSF) and blood was collected, during the first 3 weeks, then prepared for storage and later analyzed. Samples were stored in -70 degrees Celsius until analyzed. 1 year after trauma patients were assessed according to Glasgow outcome scale (GOS), NIHSS and Barthels Index. 10-15 years after trauma an evaluation of GOS by phone was repeated. Biomarkers such as Neurofilament light, Glial fibrillary acidic protein, Tau among others is analyzed in serum and CSF. Further, patients APOE genotype was explored. The investigators hypothesizes that higher concentrations of these biomarkers both in serum and CSF relate to worse 1-year and 10-15 year outcome after a severe traumatic brain injury. Further, patients that have the gene APOE4 is predisposed to worse 1 year and 10-15 year outcome after a sTBI. The investigators further want to explore the dynamics of these biomarkers in serum and CSF in the acute phase after trauma and if these biomarkers gave any prognostic value to on outcome (mortality and functional) 1-year and 10-15 years after trauma.

ELIGIBILITY:
Inclusion Criteria:

* Reaction level scale >3, corresponding to a Glasgow coma scale <9
* A therapeutic indication for intracranial pressure monitoring
* Need for ventilator treatment

Exclusion Criteria:

* Not residing in Sweden

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with severe traumatic brain injury, defined by our inclusion criteria, where enrolled from the Neurointensive care unit at Sahlgrenska university hospital, Gothenburg. Sahlgrenska University hospital is a tertiary hospital admitting patients from the whole south west part of Sweden.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2000-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
In severe traumatic brain injury patient; Correlation of Neurochemical biomarkers analyzed in CSF and serum, assessed in the initial ICU period, correlated to Glasgow Outcome Scale (GOS) at 1 year post-trauma | 1 year after trauma
  GOS 1-3 - Poor outcome, GOS 4-5 Good outcome
In severe traumatic brain injury patient; Correlation of Neurochemical biomarkers analyzed in CSF and serum, assessed in the initial ICU period, correlated to Glasgow Outcome Scale (GOS) at 10-15 years post-trauma | 10-15 years after trauma
  GOS 1-3 - Poor outcome, GOS 4-5 Good outcome
In severe traumatic brain injury patient; correlation of the genetic alleles of APOE correlated to Glasgow Outcome Scale (GOS) at 1-year post-trauma) | 1 year after trauma
  GOS 1-3 - Poor outcome, GOS 4-5 Good outcome
In severe traumatic brain injury patient; correlation of the genetic alleles of APOE correlated to Glasgow Outcome Scale (GOS) at 10-15 years post-trauma) | 10-15 years after trauma
  GOS 1-3 - Poor outcome, GOS 4-5 Good outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Nellgård, MD PhD Professor, Study Director — University of Gothenburg and Västra götaland Regionen, Sahlgrenska Universitetssjukhus Mölndal
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Västra Götaland County, Sweden